CLINICAL TRIAL: NCT06198517
Title: Clinical Study of Moxibustion for the Prevention of Hemorrhagic Cystitis After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Moxibustion for the Prevention of Hemorrhagic Cystitis After Allo-HSCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Zhang (Other)
Collaborators: The First People's Hospital of Yunnan (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor-Investigator, Yi Zhang, Physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UHCT230700
Record Dates: First submitted 2023-12-21; First posted 2024-01-10 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Moxibustion; Hematopoietic Stem Cell Transplantation; Hemorrhagic Cystitis; Prevention
MeSH Terms: conditions — Cystitis, Hemorrhagic | interventions — Moxibustion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moxibustion (Experimental)
  Interventions: Other: Moxibustion
- Control (Active Comparator)
  Interventions: Other: Symptomatic treatment

INTERVENTIONS:
Other: Moxibustion — The experimental group received moxibustion of Zhongji, Guanyuan, and Qihai for 30 min qd starting on the first day after HSCT was performed until the 14th day after transplantation, while treated conventionally.
  Arms: Moxibustion
Other: Symptomatic treatment — The control group received conventional symptomatic treatment.
  Arms: Control

SUMMARY:
This study was a prospective, multicenter, randomized controlled clinical study planned to recruit 266 hematological patients with allogeneic hematopoietic stem cell transplantation (allo-HSCT), who were randomly divided into two groups according to gender, type of transplantation, and type of primary disease. The control group was treated conventionally, and the experimental group increased moxibustion of Zhongji, Guanyuan and Qihai for 30 min qd starting on the first day after HSCT was performed until the 14th day after transplantation. Urine routine tests were performed at the time of admission, +1d, and +14d, and urine BK virus, JC virus, and adenovirus were tested at four time points, namely, +1d, +14 days, onset of hematuria symptoms, and remission of HC, respectively; routine urine tests were performed once every 7 days for all patients within 100days. For patients with Hemorrhagic cystitis (HC), daily severity grading, pain scoring, cystitis symptom scoring, use of antispasmodic and analgesic medications, and major TCM evidence were recorded with the aim of evaluating the efficacy of moxibustion in the prevention of HC in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are fully aware of the study, participate voluntarily and sign the informed consent form (ICF);
2. Age: 14-60 years;
3. Patients with pernicious blood diseases undergoing allo-HSCT using the MAC protocol or patients with severe aplastic anemia (Severe aplastic anemia; severeaplasticanimin, SAA) undergoing allo-HSCT;

Exclusion Criteria:

1. refuse to participate in this clinical study;
2. The corresponding skin at the moxibustion site is broken or sensitive;
3. allo-HSCT pretreated with the RIC program;

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 266 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
highest pain score in HC patients within 100 days of transplantation | 100 days
  highest pain score in HC patients within 100 days of transplantation

SECONDARY OUTCOMES:
Weighted Pain Score (WPS) in HC within 100 days post-transplant | 100 days
  Weighted Pain Score (WPS) is a method used to assess the overall pain burden by considering both the intensity and the duration of pain. Steps to Calculate WPS:
  Record Pain Intensity : Measure the patient's pain at various time points during the study or treatment.
  Determine Time Intervals : Record the duration for which the pain was experienced at each time point.
  Assign Weights : Weights are typically assigned based on the clinical significance of the time period. For example, if a patient experiences severe pain for a prolonged period, that period would have a higher weight.
  Calculate the WPS: Multiply the pain intensity by the duration and the weight for each time period, and sum all these values to get the total WPS.
incidence of HC within 100 days post-transplant | 100 days
Granulocyte implantation rate | 100 days
Platelet implantation rate | 100 days
Incidence of acute graft-versus-host disease | 100 days
Cytomegalovirus (CMV)/Epstein-Barr virus (EBV) reactivation | 100 days
Infection | 100 days
No relapse mortality, NRM | 100 days

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Department of Hematology, The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Zhengzhou, Henan
  - Yi Zhang, Wuhan, Hubei
  - Hematology Department, The First People's Hospital of Yunnan, Kunming, Yunnan
  - Bone Marrow Transplantation Center, The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang AK, Foca MD, Jin Z, Vasudev R, Laird M, Schwartz S, Qureshi M, Kolb M, Levinson A, Bhatia M, Kung A, Garvin J, George D, Della-Latta P, Whittier S, Saiman L, Satwani P. Bacterial bloodstream infections in pediatric allogeneic hematopoietic stem cell recipients before and after implementation of a central line-associated bloodstream infection protocol: A single-center experience. Am J Infect Control. 2016 Dec 1;44(12):1650-1655. doi: 10.1016/j.ajic.2016.04.229. Epub 2016 Jul 1. PMID 27378008
- [Background] Mackall C, Fry T, Gress R, Peggs K, Storek J, Toubert A; Center for International Blood and Marrow Transplant Research (CIBMTR); National Marrow Donor Program (NMDP); European Blood and Marrow Transplant Group (EBMT); American Society of Blood and Marrow Transplantation (ASBMT); Canadian Blood and Marrow Transplant Group (CBMTG); Infectious Disease Society of America (IDSA); Society for Healthcare Epidemiology of America (SHEA); Association of Medical Microbiology and Infectious Diseases Canada (AMMI); Centers for Disease Control and Prevention (CDC). Background to hematopoietic cell transplantation, including post transplant immune recovery. Bone Marrow Transplant. 2009 Oct;44(8):457-62. doi: 10.1038/bmt.2009.255. No abstract available. PMID 19861978
- [Background] Gutierrez-Aguirre CH, Esparza-Sandoval AC, Palomares-Leal A, Jaime-Perez JC, Gomez-Almaguer D, Cantu-Rodriguez OG. Outpatient haploidentical hematopoietic stem cell transplant using post-transplant cyclophosphamide and incidence of hemorrhagic cystitis. Hematol Transfus Cell Ther. 2022 Apr-Jun;44(2):163-168. doi: 10.1016/j.htct.2020.09.149. Epub 2020 Dec 4. PMID 33814347
- [Background] Dalianis T, Ljungman P. Full myeloablative conditioning and an unrelated HLA mismatched donor increase the risk for BK virus-positive hemorrhagic cystitis in allogeneic hematopoetic stem cell transplanted patients. Anticancer Res. 2011 Mar;31(3):939-44. PMID 21498717
- [Background] Manikandan R, Kumar S, Dorairajan LN. Hemorrhagic cystitis: A challenge to the urologist. Indian J Urol. 2010 Apr;26(2):159-66. doi: 10.4103/0970-1591.65380. PMID 20877590
- [Background] Khojasteh NH, Zakerinia M, Ramzi M, Haghshenas M. A new regimen of MESNA (2-mercaptoethanesulfonate) effectively prevents cyclophosphamide-induced hemorrhagic cystitis in bone marrow transplant recipients. Transplant Proc. 2000 May;32(3):596. doi: 10.1016/s0041-1345(00)00906-4. No abstract available. PMID 10812128
- [Background] Arango M, Cardona D. Hemorrhagic Cystitis after Haploidentical Transplantation with Post-Transplantation Cyclophosphamide: Protective Effect of MESNA Continuous Infusion. Biol Blood Marrow Transplant. 2020 Aug;26(8):1492-1496. doi: 10.1016/j.bbmt.2020.04.028. Epub 2020 May 15. PMID 32417488
- [Background] Visintini C, Venturini M, Palese A. Haemorrhagic cystitis, preventive and treatment interventions in patients undergoing haematopoietic stem cell transplantation: A scoping review. Eur J Oncol Nurs. 2019 Oct;42:50-62. doi: 10.1016/j.ejon.2019.07.005. Epub 2019 Jul 12. PMID 31446264